CLINICAL TRIAL: NCT05301114
Title: Scaling Social Determinants of Health Screening, Social Support, and Anti-Racism Training to Reduce Inequities in Minority Cancer Survivor Health and Well-Being in Washington, D.C.
Brief Title: Social Risk Factors and Discrimination in Cancer Survivorship
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Collaborators: George Washington University (Other); Howard University (Other); Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 4397
Record Dates: First submitted 2022-03-16; First posted 2022-03-29 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-05

CONDITIONS: Social Determinants of Health; Breast Cancer; Prostate Cancer; Health Equity; Disparities
Keywords: Health Equity; Community Health Worker; Social Support; Community Based Organizations; Social Determinants of Health; Breast Cancer; Prostate Cancer; Health Disparities
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention participants (Experimental): Among patients who completed the social needs screening as a part of standard of care, all stage I-IV Black cancer survivors will be invited to participate in a six-month community health worker intervention. The community health worker will assess social needs and provide six months of support.
  Interventions: Behavioral: Community Health Worker support

INTERVENTIONS:
Behavioral: Community Health Worker support — Participant will receive weekly or monthly support (via phone or in person) from a community health worker. The community health worker will be responsible for continuously assessing the patient's social needs, providing referrals to community based organizations, and assisting with the patient's non-medical needs as they progress through survivorship (e.g. social support, referrals, etc). Individuals who identify no risk factor will receive monthly phone calls, while individuals who identify 1-3 risk factors will receive monthly home visits with interim phone calls for 6 months. Those who identify 4 or more risk factors or have intensive needs such as behavioral health will receive the same services as the medium risk group and will also be connected with the social work teams within each institution.

SUMMARY:
The objective of the proposed study is to scale social risk factor screening and referral for cancer survivors and to solidify information exchange between clinical and community settings in order to improve survivor health and well-being. This will be completed through three primary aims: 1) To ascertain workflow and map community resources needed to facilitate social risk factor screening and referral for breast and prostate cancer survivors in Washington, District of Columbia. 2) To determine impact of Community Health Worker (CHW) support on Black breast and prostate cancer survivor health and wellbeing as measured through quality of life (QOL) and social connection. 3) To determine impact of anti-racism training for staff and clinicians at three cancer centers on patient-reported discrimination.

DETAILED DESCRIPTION:
Despite improvements in cancer outcomes over time, significant disparities remain between Black and White cancer survivors. It is estimated that clinical care, including access to care and quality of care, accounts for an estimated 20% of health outcomes, while other factors, including social determinants of health (SDoH) and an individual's social risk factors, explain 80% of health outcomes. The goal of this research is thus to simultaneously target unequitable health care systems and accelerate the evidence base for scalable social determinants of health screening and referral to reduce inequities in cancer survivor health and well-being. This project is intended to establish sustainable clinical-community linkages and improve survivor health and well-being. Understanding the burden of social needs in this population, the available community resources, and solidifying integrated, closed-loop referral systems to address those needs is critical to improving quality of life for cancer survivors. The long-term goal of this research is to develop scalable interventions to address social needs and support for cancer survivors.

The study aims to: 1) improve care coordination and information exchange through mapping available resources for cancer survivors across Washington DC and building a universal screening and referral process at three cancer centers in DC; 2) determine impact of Community Health Worker (CHWs) support on cancer survivor health and wellbeing as measured through social connection and quality of life; 3) determine impact of anti-racism (inclusive of SDOH) training for staff and clinicians at three cancer centers on provider cultural competency and patient reported perceived discrimination.

Furthermore, this work evaluates the implementation, impact, and causal mechanisms of SDOH collection and referral to reduce racial inequities among cancer survivors. The investigators include innovative approaches to linking clinics and communities drawing on systems engineering and social network analyses and supported by ongoing DC efforts to bolster health information exchange systems to address social needs. Our approach is also integrated with existing community resources including key community-based organizations in the Washington DC region.

Results from this study will provide the foundation for future research examining the intervention's generalizability to other marginalized cancer survivors and sustainability of the proposed screening and referral system. Findings will also provide a basis for further research on community health workers to support our target population, to improve shared resources in supporting cancer survivors, and to maintain relevance within the evolving health information exchange environment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stage I-III breast or prostate cancer and completed curative treatment (surgery, radiation, chemotherapy) or finalized treatment plan (e.g. watch and wait); OR Stage IV breast or prostate cancer approximately 6 months from diagnosis
* Black or African American race

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1116 (Estimated)
Dates: Start 2022-05-05 (Actual); Primary Completion 2026-07-20 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Patient Self-Efficacy | 6 months
  This study will use the following Patient-Reported Outcomes Measurement Information System® (PROMIS) self-efficacy for managing chronic conditions 4-item measures: managing daily activities, managing emotions, managing medications and treatments, and managing social interactions. The minimum score on these overall scales is a 16 and the maximum score is 80, in which a higher number represents a higher level of self-efficacy for managing chronic conditions. PROMIS raw scores are then transformed to a t-scale with a mean of 50 and a standard deviation of 10.
Health-related quality of life (QOL) | 6 months
  QOL will be measured using the Patient-Reported Outcomes Measurement Information System® (PROMIS) 29 computer adaptive test, a collection of 4-item adaptive forms assessing physical function, anxiety, depression, fatigue, sleep disturbance, ability to participate in social roles and activities, pain interference, as well as a single global pain item. For the 4-item forms, the lowest score is 4 and the highest score is 16. Higher scores represent higher levels of physical function, anxiety, depression, fatigue, sleep disturbance, ability to participate in social roles and activities, pain interference, respectively. The single pain item has a minimum score of 0 and a maximum score of 10, in which a higher score represents a higher level of pain. PROMIS raw scores are then transformed to a t-scale with a mean of 50 and a standard deviation of 10.
Social connectedness | 6 months
  To measure social connectedness, this study will draw from the item banks for the following Patient-Reported Outcomes Measurement Information System® (PROMIS) 2.0 adult item measures: Social Isolation, Emotional Support, Informational Support, and Instrumental Support. Each scale is scored with a minimum score of 4 and a maximum score of 20, in which higher scores represent higher levels of social isolation, emotional support, instrumental support, and informational support, respectively. PROMIS raw scores are then transformed to a t-scale with a mean of 50 and a standard deviation of 10.
Acceptability of the CHW intervention | 12 months
  A four-item Likert scale will be delivered to relevant clinicians to provide feedback on acceptability of the intervention
Appropriateness of the CHW intervention | 12 months
  A four-item Likert scale will be delivered to relevant providers to provide feedback on appropriateness of the intervention, whereby higher scores indicate greater perceived appropriateness.
Feasibility of the CHW intervention | 12 months
  A four-item Likert scale will be delivered to relevant providers to provide feedback on feasibility of the intervention, whereby higher scores indicate greater perceived feasibility.
Sustainability Assessment | 12 months
  This study will use the Program Sustainability Assessment Tool annually to assess environmental support, funding stability, partnerships, organizational capacity, program evaluation, program adaptation, communications and strategic planning. The minimum score for this evaluation is 0 and the maximum score is 56. A higher score represents a higher level of program sustainability. Individual categories can also be assessed with a minimum score of 0 and a maximum score of 7 in each, in which a higher score represents higher sustainability in that category.

SECONDARY OUTCOMES:
Social risk factors | 3 months
  Social risk factors screeners will be administered on the following domains: food insecurity, housing instability, utilities, paying for the basics, employment, transportation, and mental health. These scales are measured uniquely to the electronic health record systems in which they are implemented. Each need is assigned a single point and summed for an overall score.

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Arem, PhD, Principal Investigator — Medstar Health Research Institute; Mandi Pratt-Chapman, PhD, Principal Investigator — George Washington University
Locations (1):
- MedStar Washington Hospital Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Glasgow RE, Kwan BM, Matlock DD. Realizing the full potential of precision health: The need to include patient-reported health behavior, mental health, social determinants, and patient preferences data. J Clin Transl Sci. 2018 Jun;2(3):183-185. doi: 10.1017/cts.2018.31. Epub 2018 Sep 13. PMID 30370072
- [Background] Clarke TC, Christ SL, Soler-Vila H, Lee DJ, Arheart KL, Prado G, Caban-Martinez A, Fleming LE. Working with cancer: health and employment among cancer survivors. Ann Epidemiol. 2015 Nov;25(11):832-8. doi: 10.1016/j.annepidem.2015.07.011. Epub 2015 Aug 4. PMID 26320705
- [Background] Weaver KE, Rowland JH, Bellizzi KM, Aziz NM. Forgoing medical care because of cost: assessing disparities in healthcare access among cancer survivors living in the United States. Cancer. 2010 Jul 15;116(14):3493-504. doi: 10.1002/cncr.25209. PMID 20549763
- [Background] Cella D, Yount S, Rothrock N, Gershon R, Cook K, Reeve B, Ader D, Fries JF, Bruce B, Rose M; PROMIS Cooperative Group. The Patient-Reported Outcomes Measurement Information System (PROMIS): progress of an NIH Roadmap cooperative group during its first two years. Med Care. 2007 May;45(5 Suppl 1):S3-S11. doi: 10.1097/01.mlr.0000258615.42478.55. PMID 17443116
- [Background] Cella D, Riley W, Stone A, Rothrock N, Reeve B, Yount S, Amtmann D, Bode R, Buysse D, Choi S, Cook K, Devellis R, DeWalt D, Fries JF, Gershon R, Hahn EA, Lai JS, Pilkonis P, Revicki D, Rose M, Weinfurt K, Hays R; PROMIS Cooperative Group. The Patient-Reported Outcomes Measurement Information System (PROMIS) developed and tested its first wave of adult self-reported health outcome item banks: 2005-2008. J Clin Epidemiol. 2010 Nov;63(11):1179-94. doi: 10.1016/j.jclinepi.2010.04.011. Epub 2010 Aug 4. PMID 20685078
- [Background] Hahn EA, Devellis RF, Bode RK, Garcia SF, Castel LD, Eisen SV, Bosworth HB, Heinemann AW, Rothrock N, Cella D; PROMIS Cooperative Group. Measuring social health in the patient-reported outcomes measurement information system (PROMIS): item bank development and testing. Qual Life Res. 2010 Sep;19(7):1035-44. doi: 10.1007/s11136-010-9654-0. Epub 2010 Apr 25. PMID 20419503